CLINICAL TRIAL: NCT03902067
Title: Safety and Efficacy Evaluation of Umbilical Cord Mesenchymal Stem Cells Transcatheter Transplantation to Treat Left Ventricular Dysfunction After Acute Myocardial Infarction
Brief Title: UC-MSC Transplantation for Left Ventricular Dysfunction After AMI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Life Science & Technology (Industry)
Collaborators: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiLST-ucmsc-ami01
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2023-10

CONDITIONS: Left Ventricular Dysfunction; Acute Myocardial Infarction
Keywords: AMI
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UC-MSC (Experimental): UC-MSC transplantation
  Interventions: Biological: UC-MSC
- Control Group (Placebo Comparator): Routine treatment
  Interventions: Biological: Control Group

INTERVENTIONS:
Biological: UC-MSC — 0.25ml Shanghai Life UC-MSC injection is resuspended into 10ml of cell suspension and slowly infused into infarct-related blood vessels through an administration catheter in 2 minutes, and the number of cells transplanted each time is 5x10(6) cells. The UC-MSC products are manufactured by Shanghai Life with viability>80%, and endotoxin<0.1 EU， at the concentration of 2x10(7) cells/ml.
  Other Names: Transplantation Group
  Arms: UC-MSC
Biological: Control Group — Routine treatment without catheter infusion
  Arms: Control Group

SUMMARY:
A pilot study to evaluate the safety and feasibility of umbilical cord mesenchymal stem cells in the treatment of acute myocardial infarction by catheter transplantation

DETAILED DESCRIPTION:
In this study, 40 patients with cardiac insufficiency after acute myocardial infarction were selected and randomly divided into umbilical cord MSCs transplantation treatment group and non-intervention control group to preliminarily observe the safety and effectiveness of MSCs cell transplantation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute extensive anterior myocardial infarction were successfully treated with emergency interventional therapy within 12 hours after onset. LVEF was less than 0.35 by echocardiography 30 days after operation, scar area was more than 25% by MRI, and cardiac function was NYHA III-IV grade.
* Fully inform the purpose, method and possible side effects of the test, agree to the test, and sign an informed consent form;
* Good compliance, willing to take drugs and follow up according to the requirements of the plan;
* Life expectancy exceeds one year.

Exclusion Criteria:

* Those who cannot tolerate cell therapy;
* Patients with severe hepatic and renal insufficiency (ALT>1.5 times the upper limit of normal value, Cr >1.5 times the upper limit of normal value);
* Patients with malignant tumors or extremely weak patients;
* Patients with severe infection;
* Patients who are expected to have the second coronary intervention or bypass grafting within 3 months;
* Patients with other serious systemic diseases and organ dysfunction;
* Patients with cardiogenic shock;
* Patients with hemorrhagic diseases;
* Researchers believe that anyone who is not suitable for inclusion

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety measured as the number of Major Adverse Cardiac Events (MACE) | 12 months
  Possible adverse events, including adverse events that may occur during angiography and infusion of transplanted cells such as chest pain, arrhythmia, slow blood flow, myocardial injury, fever, allergic reaction, postoperative infection, etc.

SECONDARY OUTCOMES:
Difference in left ventricular ejection fraction measured by magnetic resonance imaging at baseline and 12 months follow-up | 12 months
  left ventricular ejection fraction measured by magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Chengxing Shen, Dr., Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (1):
- Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, Shanghai Municipality, China